CLINICAL TRIAL: NCT05068921
Title: Phase I Clinical Trial to Evaluate Tolerability and Pharmacokinetics of TQB2858 Injection in Subjects With Advanced Malignancy
Brief Title: A Clinical Trial to Evaluate Tolerability and Pharmacokinetics of TQB2858 Injection in Subjects With Advanced Malignancy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-Ⅰ-06
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Advanced Cervical Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 (Experimental): TQB2858 injection: once every 3 weeks, 1800mg each time, intravenous infusion. Until the disease progression or unbearable adverse events occur.
  Interventions: Drug: TQB2858 injection

INTERVENTIONS:
Drug: TQB2858 injection — TQB2858 is an anti-programmed death ligand 1（PD-L1）/transforming growth factor-β （TGF-β） bi-functional fusion protein.

SUMMARY:
A phase I clinical trial of tolerability and pharmacokinetics of TQB2858 injection in subjects with advanced malignancy.

ELIGIBILITY:
Inclusion Criteria:

* 1) All the following conditions were met for the corresponding study stage:

  a) Cervical cancer confirmed by histopathology, including squamous carcinoma, adenocarcinoma and adenosquamous carcinoma; b) Have received ≥1 line of platinum-containing chemotherapy (at least ≥3 cycles of platinum-containing chemotherapy) in the past, and have disease progression or recurrence during or after treatment; c) Confirmed presence of at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 standard;
* 2) Aged: 18 ~ 75 years old
* 3)Physical condition score( Eastern Cooperative Oncology Group(ECOG) score): 0~1
* 4) estimated survival time ≥ 3 months
* 5)The main organs function well and meet the following standards:

  a) Routine blood examination standards (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days before screening):Hemoglobin (HGB) ≥80 g/L; Neutrophil count (NEUT) ≥ 1.5×109/L; Platelets (PLT)≥90×109 /L; b) Biochemical examination: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (Primary hepatobiliary tumor or liver metastasis: ALT, AST≤ 5×ULN ); Total bilirubin (TBIL) ≤1.5×ULN (Gilbert syndrome patients: TBIL≤ 3×ULN); Creatinine (CRE) ≤ 1.5×ULN or creatinine clearance ≥ 60 mL /min; c) Blood coagulation function: activated partial thrombin time (APTT), international standardized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN (without anticoagulant therapy); d) Left ventricular ejection fraction (LVEF) ≥ 50%;
* 6) Female subjects of childbearing age should agree to use effective contraceptive measures (such as intrauterine device , birth control pills or condoms) during the study period and within 6 months after the end of the study, and have a negative serum pregnancy test within 7 days before the study enrollment and must be non-lactating subjects;
* 7）The subjects voluntarily joined the study, signed the informed consent form, and had good compliance.

Exclusion Criteria:

* 1) Combined following diseases or medical history:

  1. the presence of other malignant tumors within 2 years or current co-occurrence . The following two conditions can be included: other malignant tumors treated by single surgery, achieved R0 resection and no recurrence and metastasis; Cured cervical carcinoma in situ (only applicable to the first stage), non-melanoma skin cancer, nasopharyngeal carcinoma, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basal membrane)];
  2. Pathological findings of mucinous adenocarcinoma, clear cell adenocarcinoma, neuroendocrine tumor and other special pathological types (only applicable to the second stage);
  3. Evaluation criteria for common adverse events(CTCAE) grade> 1 unrelieved toxicity of due to any prior treatment, excluding hair loss and peripheral sensory nerve disorders;
  4. major surgical treatment or significant traumatic injury within 28 days prior to the start of study treatment (excluding needle aspiration, endoscopic biopsy for diagnostic purposes, etc.);
  5. wounds or fractures that have not been cured for a long time;
  6. Occurrence of arteriovenous/venous thrombosis events within 6 months, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
  7. those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
  8. Subject with any severe and/or uncontrolled disease, including:

     1. Patients with poor blood pressure control after standard treatment (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥ 100mmHg);
     2. Patients who have experienced myocardial ischemia or myocardial infarction within six months; New York Heart Association(NYHA )grade ≥2 congestive heart failure; Grade ≥2 atrioventricular block; Arrhythmias that cannot be stably controlled with drugs (including QTc ≥470ms) and arrhythmias that may have a potential impact on trial treatment;
     3. Active infection ( CTCAE grade ≥ 2 infection);
     4. Decompensated liver cirrhosis, active hepatitis *;

        * active hepatitis (hepatitis B reference:Hepatitis B surface antigen( HBsAg )positive, and Hepatitis B virus DNA(HBV DNA)>2500 copies /mL or > 500 IU/mL; Hepatitis C reference: hepatitis C virus(HCV) antibody positive, and HCV virus titer test value exceeds the upper limit of normal value); Note: Subjects with positive surface antigen of hepatitis B or positive core antibody and hepatitis C patients eligible for inclusion are advised to continue antiviral therapy to prevent virus activation;
     5. Active syphilis and active tuberculosis;
     6. Renal failure requiring hemodialysis or peritoneal dialysis: glomerular filtration rate(eGFR) < 15ml/ (min•1.73㎡);
     7. A history of immunodeficiency, including Human Immunodeficiency Virus(HIV )positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation;
     8. Poor control of diabetes (Fasting blood glucose (FBG) > 10mmol/L, bedtime blood glucose > 11.1mmol/L and hemoglobin A1C (HbA1c) ≥8.5% before bedtime);
     9. Patients with urine protein ≥++ as indicated by routine urine examination, and 24-hour urine protein quantity > 1.0g;
     10. Persons suffering from epilepsy and requiring medical treatment.
* 2) Tumor-related symptoms and treatment: a) Received surgery, chemotherapy, radiation or other anticancer therapy within 4 weeks before the start of study treatment (the washout period is calculated from the end of the last treatment); Those who had previously received local radiation therapy were eligible to enroll if they met the following criteria: the end of radiotherapy was more than 4 weeks before the start of study therapy (brain radiation was more than 2 weeks); The target lesions selected in this study are not in the radiotherapy region. Or the target lesion is located in the radiotherapy area, but progression is confirmed. b) Received the treatment of Chinese patent medicines with anti-tumor indications specified in the National Medical Products Administration(NMPA) approved drug instructions (including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.) within 2 weeks before the study treatment; c) Previously received immunomodulator therapy, including therapeutic vaccines, cytokine therapy, or Anti-programmed death receptor 1(anti-PD-1), Programmed death ligand-1(PD-L1), Cytotoxic T lymphocyte-associated protein 4(CTLA-4), High purity recombinant protein(4-1BB), T cell activation markers(OX-40) and other related immunotherapy drugs; d) pleural effusion, pericardial effusion, or ascites that uncontrolled and still requires repeated drainage (as determined by the investigator); e) Patients with brain metastasis whose symptom control stabilizes for less than 4 weeks after withdrawal of dehydrants and steroids (only for stage 2 patients with previous central nervous system metastases).
* 3) Research treatment related: a) history of live attenuated vaccine administration within 28 days before the start of study treatment or planned live attenuated vaccine administration during the study period; b) Have a history of severe allergy to macromolecule drugs or known components of TQB2858 injection; c) An active autoimmune disease requiring systemic treatment (such as palliative drugs, corticosteroids, or immunosuppressants) occurred within 2 years before the start of study therapy. Alternative therapies (such as thyroxine, insulin, or physical corticosteroids for adrenal or pituitary dysfunction, etc.) are not considered systemic treatment; d) diagnosed as immunodeficient or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose >10mg/ d of prednisone or other equivalent hormone) and continued use within 2 weeks of initial administration; e) Participated in clinical trials of other antitumor drugs within 4 weeks before grouping.
* 4) According to the researcher's judgment, subjects who have concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or who are considered unsuitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | Baseline to up to two years
  Proportion of patients whose tumors shrank by a certain amount and remained for a certain period of time, including complete response (CR) and partial response (PR) .

SECONDARY OUTCOMES:
Progress Free Survival(PFS) | Baseline to up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first)
Disease Control Rate(DCR) | Baseline to up to two years
  Proportion of subjects whose tumors shrink or remain stable for a certain period, including complete remission（CR）, partial remission（PR） and stable disease（SD）
Duration of Response(DOR) | Baseline to up to two years
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first) .
Overall Survival(OS) | Baseline to up to two years
  The period from the first use of the drug to death from all causes. For subjects who are still alive at the last follow-up, the OS will be counted as data censored based on the last follow-up. For subjects who are lost follow-up, the OS will be counted as data censored based on the last confirmed survival time before being lost to follow-up.
Occurrence of all adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs) | Baseline to up to two years
  Adverse events refer to all adverse medical events that occur after a patient or clinical trial subject receives an experimental drug, which can be expressed as symptoms, signs, diseases, or abnormalities in laboratory tests, but are not necessarily related to the treatment of the experimental drug. Serious adverse events refer to adverse medical conditions such as death, life threatening, permanent or severe disability, loss of function, the need for hospitalization or prolonged hospitalization , and congenital abnormalities or birth defects after the subject receives the experimental drug.

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Third Affiliated Hospital of Qiqihar Medical College, Qiqihar, Heilongjiang
  - Hunan Cancer Hospita, Changsha, Hunan
  - Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Linyi Tumor Hospital, Linyi, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Affiliated Peace Hospital of Changzhi Medical College, Changzhi, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xian, Shanxi
  - Sichuan Cancer Hospita, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality